CLINICAL TRIAL: NCT03604601
Title: Analysis of the Curative Effect of Salvage Surgery on Recurrent Laryngeal Carcinoma: A Single-institutional Experience
Brief Title: Analysis of the Curative Effect of Salvage Surgery on Recurrent Laryngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, GengLong Liu, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: recurrent laryngeal carcinoma
Record Dates: First submitted 2018-07-13; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Laryngeal Carcinoma
Keywords: salvage surgery; recurrent laryngeal carcinoma; experience
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: salvage surgery — Salvage surgery hopes to control the recurrence of larynx, pharynx, fistula and neck tumor and improve the quality of life and survival rate

SUMMARY:
Early laryngeal cancer can be treatment by laser surgery or radiotherapy, intermediate and advanced laryngeal carcinoma mainly surgical treatment. Laryngeal cancer is at risk of recurrence after treatment, whether in surgery, laser or radiotherapy. The recurrence rate of laryngeal cancer is about 10% reported at home and abroad. Local pain, ulcers, breathing and eating difficulties caused by recurrent laryngeal cancer seriously reduce the quality of life of patients and seriously endanger their lives. Therefore, head and neck surgeons are required to make every effort to give them saving treatment in order to improve their quality of life. Prolong the patient's life.

DETAILED DESCRIPTION:
medical records and extracted information including age, gender, initial treatment modality of glottis cancer, recurrence time, recurrence site, histopathology, tumor grade according to World Health Organization (WHO) grade and tumor stage. Stages were defined according to the American Joint Committee on Cancer (AJCC) staging system.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years,
* patients with recurrent glottic laryngeal squamous cell carcinoma undergoing salvage surgery

Exclusion Criteria:

* postoperative radiotherapy and chemotherapy
* loss to follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with recurrent laryngeal squamous cell carcinoma
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | Follow up 5 years
  The overall survival rate was calculated with Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Genglong Liu, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Undecided